CLINICAL TRIAL: NCT01502189
Title: Information to Parents of Children With Cancer. An Exploratory Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Ulla Hallgren Graneheim, Associate professor, Umeå University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PROJ07/029
Record Dates: First submitted 2011-12-21; First posted 2011-12-30 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Stress; Health Knowledge, Attitudes, Practice
Keywords: patient education as topic; representational approach; parents; childhood cancer; paediatric oncology; nursing; parents of children with cancer; Stress; Health Knowledge; Attitudes; Practice
MeSH Terms: conditions — Behavior; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Representational approach (Experimental): The Representational approach as described in the detailed description.
  Interventions: Other: Representational approach

INTERVENTIONS:
Other: Representational approach — The Representational approach as described in the detailed description. Each participating parent receives three rounds that consist of two meetings. Each round starts with a meeting where the parent identifies an area where he/she needs more information. The nurse and the parent jointly survey the parent's representation of the area and discusses consequences of knowledge gaps or misunderstandings. Then, new information is introduced and benefits from the new information is discussed. After some days, a follow-up meeting takes place.

SUMMARY:
The aim of this study is to explore whether an intensified informational intervention built upon the Representational approach framework can reduce stress in parents of children with cancer.

DETAILED DESCRIPTION:
BACKGROUND

Parents of children with cancer have great information needs and report that these are not always met. Psychosocial suffering such as stress and anxiety is also common in this group.

HYPOTHESIS

An informational intervention emanating from the needs identified by parents is associated to decreased perceived stress, decreased depressive symptoms, decreased anxiety, increased satisfaction with information and decreased use of health care contacts in parents.

INTERVENTION

The intervention builds upon the Representational approach. This approach emanates from Leventhal's theories of illness representations and theories of conceptual change. Central qualities in the approach is that parents identify the area where information is needed themselves and that a thorough assessment of their current representation of that area is performed before information is given.

Each participating parent receives three rounds that consist of two meetings. Each round starts with a meeting where the parent identifies an area where he/she needs more information. The nurse and the parent jointly survey the parent's representation of the area and discusses consequences of knowledge gaps or misunderstandings. Then, new information is introduced and benefits from the new information is discussed. After some days, a follow-up meeting takes place.

DESIGN AND METHODS

The intervention will be evaluated using a single-case design (A-B-A-B-A-B-A) with 10 parents. All parents will receive the intervention, and repeated measures of the outcome variables both before and after will be used to assess the effect of the intervention. Data will be collected by web questionnaires with SMS- and e-mail reminders.

In parallel, a process evaluation aiming at describing treatment fidelity, experiences of participation and impact of contextual factors on the results. For this aim, qualitative interviews with participants and audio recording of intervention sessions will be used.

ELIGIBILITY:
Inclusion Criteria:

* Being a parent of a child that

  1. is diagnosed with a first occurrence of a malignancy that is curatively treated
  2. was diagnosed two months ago
* Able to talk, read and write Swedish enough to be able to participate without an interpreter
* Have access to a computer and an internet connection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Perceived stress | Changes during baseline and intervention period (measured twice a week for a total of 11 weeks).
  As measured by the Perceived stress scale (PSS). 10 items answered on a 5-point Likert scale.

SECONDARY OUTCOMES:
Physical symptoms from stress | Changes during baseline and intervention period (measured twice a week for a total of 11 weeks).
  Includes headache, sleep disturbances, palpitations, and heartburn, each measured on a 4-point scale.
Anxiety | Changes during baseline and intervention period (measured twice a week for a total of 11 weeks).
  Measured on a 7-point visual digital scale.
Depressive symptoms | Changes during baseline and intervention period (measured twice a week for a total of 11 weeks).
  Measured on a 7-point visual digital scale.
Satisfaction with information | Changes during baseline and intervention period (measured twice a week for a total of 11 weeks).
  Includes general satisfaction with the information from the health care professionals as well as information from the intervention nurses. Measured on a 7-point visual digital scale.
Healthcare contacts | Changes during baseline and intervention period (measured once a week for a total of 11 weeks).
  Number of contacts with the health care system concerning the ill child and the parent's own health problems.

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Hällgren Graneheim, Associate professor, Study Director — Umeå University
Locations (1):
- Umeå University Hospital, Umeå, Västerbotten County, Sweden